CLINICAL TRIAL: NCT01635582
Title: Effects of Home Based Computer Gaming Hand Exercise Regimen in People With Rheumatoid Arthritis (RA) or Osteoarthritis (OA) -A Randomized Controlled Pilot Trial
Brief Title: Home Based Computer Gaming Hand Exercise Regimen for People With Arthritis Affecting the Hands
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Arthritis Network (Network)
Responsible Party: Principal Investigator, Dr. Tony Szturm, Associate Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H2012:182
Record Dates: First submitted 2012-06-29; First posted 2012-07-09 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis of Hands
Keywords: Hand exercises; Hand function; Computer based exercises; Therapeutic gaming
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): Conventional hand exercise program
  Interventions: Other: Conventional hand exercise program
- Experimental group (Experimental): Computer gaming hand exercise regimen'
  Interventions: Other: Computer gaming hand exercise regimen

INTERVENTIONS:
Other: Conventional hand exercise program — Exercises targeted to improve finger range of motion and hand strength.The exercises will be performed 30 minutes,four times per week for six weeks
  Arms: Control group
Other: Computer gaming hand exercise regimen — Computer gaming hand exercise regimen using common objects of daily life. The hand exercises are coupled with commercially available computer games and will be performed 30 minutes,four times per week for six weeks
  Arms: Experimental group

SUMMARY:
The purpose of the study is to determine whether a novel computer gaming hand exercise regimen would improve hand function, decrease pain/ stiffness and be feasible in people with Rheumatoid arthritis or Osteoarthritis affecting the hands.

DETAILED DESCRIPTION:
A novel computer gaming hand exercise regimen has been designed for people with Rheumatoid arthritis (RA) or Osteo arthritis (OA) affecting the hands. The design allows a broad range of common objects of daily life to be seamlessly transformed into 'therapeutic' input devices by instrumenting with a small motion sense mouse. Based on individual abilities and treatment needs, objects are selected to train specific fine/ gross dexterous functions. The object manipulations (therapeutic exercises) are then used to control and play any commercially available computer game, making practice challenging and engaging.

The study is of six weeks duration comparing the computer gaming and conventional hand exercises in thirty people diagnosed with RA or OA affecting the hands. The investigators hypothesize that the game based exercises will improve hand function and reduce pain/stiffness and be feasible compared to the conventional hand exercises.A mixed-effect repeated measures analysis of variance will be conducted to test pre to post treatment outcomes. This will be the first study to evaluate the therapeutic effects and feasibility of the computer gaming hand exercise regimen in people with RA or OA.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Aged between 30-70 years
* Clinical diagnosis of Rheumatoid arthritis or Osteoarthritis of hands according to American college of rheumatology criteria
* Must own a home computer and have basic working knowledge of computers.
* Present with scores ranging from 0-75 on self-reported hand function ability with the Disabilities of Arm, Shoulder and Hand (DASH) questionnaire

Exclusion Criteria:

* Severely deformed finger joints
* Neurological conditions of dominant side upper limb
* Trauma in wrist or hand
* Upper limb surgeries in previous six months
* Co-existing hand conditions in the dominant hand
* Problems with vision or hearing
* Recent changes in drug regimen (Disease modifying anti-rheumatic drugs (DMARDs) or corticosteroids <3 months)
* Major diseases of heart or lungs or liver
* DASH scores 0-75.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Arthritis Hand Function Test (AHFT) at 6 weeks | Baseline and 6 weeks
  The Arthritis Hand Function Test(AHFT) is an 11-item performance based test to measure grip and pinch strength, dexterity, applied strength and applied dexterity in people with arthritis.

SECONDARY OUTCOMES:
Change from baseline in Disabilities of Arm,Shoulder and Hand(DASH) questionnaire at 6 weeks | Baseline and 6 weeks
  The DASH is a self-report questionnaire, with 30 items designed to measure functional ability and symptoms in people with any of several musculo skeletal disorders of the upper limb
Change from baseline in Paddle game based hand function assessment tool at 6 weeks | Baseline and 6 weeks
  A novel, paddle game based hand function assessment tool has been developed designed to: 1) Objectively quantify the quality of finger hand movements (task performance) during manipulation of broad range of common objects independent of physical properties, anatomical requirements and task goal/context, 2) Quantify pain and joint stiffness during each object manipulation task, 3) Track changes in finger hand function over time and 4) Aid in clinical decision making
Personal exercise log diary | End of 6 weeks of home exercise program
  Exercise compliance will be measured at the end of 6 weeks of home exercise program

CONTACTS AND LOCATIONS:
Overall Officials: Tony Szturm, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Szturm T, Peters JF, Otto C, Kapadia N, Desai A. Task-specific rehabilitation of finger-hand function using interactive computer gaming. Arch Phys Med Rehabil. 2008 Nov;89(11):2213-7. doi: 10.1016/j.apmr.2008.04.021. PMID 18996252
- [Background] Lockery D, Peters JF, Ramanna S, Shay BL, Szturm T. Store-and-feedforward adaptive gaming system for hand-finger motion tracking in telerehabilitation. IEEE Trans Inf Technol Biomed. 2011 May;15(3):467-73. doi: 10.1109/TITB.2011.2125976. PMID 21536526
- [Background] Andersen Hammond ER, Shay BL, Szturm T. Objective evaluation of fine motor manipulation-a new clinical tool. J Hand Ther. 2009 Jan-Mar;22(1):28-35; quiz 36. doi: 10.1197/j.jht.2008.06.006. Epub 2008 Aug 30. PMID 18950989
- [Background] Hammond ER, Szturm T, Shay BL. Manipulation of objects with and without the use of the index finger: implications for digital amputations. J Hand Ther. 2010 Oct-Dec;23(4):352-59; quiz 360. doi: 10.1016/j.jht.2010.04.005. Epub 2010 Jul 6. PMID 20609561
- [Derived] Srikesavan CS, Shay B, Szturm T. Task-Oriented Training with Computer Games for People with Rheumatoid Arthritis or Hand Osteoarthritis: A Feasibility Randomized Controlled Trial. Games Health J. 2016 Oct;5(5):295-303. doi: 10.1089/g4h.2016.0005. Epub 2016 Sep 13. PMID 27623532
- [Derived] Srikesavan CS, Shay B, Robinson DB, Szturm T. Task-oriented training with computer gaming in people with rheumatoid arthritisor osteoarthritis of the hand: study protocol of a randomized controlled pilot trial. Trials. 2013 Mar 9;14:69. doi: 10.1186/1745-6215-14-69. PMID 23497529